CLINICAL TRIAL: NCT03750201
Title: Direct Selective Laser Trabeculoplasty (DSLT) In Open Angle Glaucoma (POAG): A Randomized Controlled Trial
Brief Title: A Study to Assess an Automated Laser Device for Direct Selective Laser Trabeculoplasty
Acronym: GLAUrious
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BelkinVision (Industry)
Collaborators: European Commission (Other); Universita degli Studi di Genova (Other); Queen's University, Belfast (Other); Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GLAUrious-2017-01
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2021-07

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Intra-ocular pressure (IOP) measurements by masked investigator or masked technique (masked reading).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct Selective Trabeculoplasty (Experimental): Treatment by the investigational device.
  Interventions: Device: Direct Selective Trabeculoplasty
- Selective Trabeculoplasty (Active Comparator): Treatment by the comparator device.
  Interventions: Device: Selective Trabeculoplasty

INTERVENTIONS:
Device: Direct Selective Trabeculoplasty — Laser surgery by automated direct automated SLT device to lower intraocular pressure
  Arms: Direct Selective Trabeculoplasty
Device: Selective Trabeculoplasty — Laser surgery by standard SLT device to lower intraocular pressure
  Arms: Selective Trabeculoplasty

SUMMARY:
Glaucoma is an eye disease that results in damage to the optic nerve that progresses over time. One of the main risk factors in glaucoma is an increase in intraocular pressure, caused by a build-up of fluid in the eye. Glaucoma can result in blindness if left untreated and as such it is extremely important to diagnose and treat the condition.

Selective Laser Trabeculoplasty (SLT) is a laser treatment that facilitates the outflow of fluid from inside the eye. This has the potential of reducing the intraocular pressure within the eye (the main way in which this disease is treated since there is no cure) and may assist in helping to control the progression of this disease.

SLT (standard treatment) is a technique routinely carried out by glaucoma specialists. It is conducted using a special type of lens (goniolens) that gently sits on the front surface of the eye. The procedure takes approximately 5 minutes in duration.

This new treatment, Direct Selective Laser Trabeculoplasty (DSLT) is performed directly, without there being any need to use a goniolens which sits on the eye, and it is a shorter and simpler technique to conduct when compared to the standard SLT technique.

The purpose of this study is to assess the hypothesis that the treatment by new automated device for DSLT is not worse in comparison with the standard SLT and determine that it is effective in reducing intraocular pressure.

DETAILED DESCRIPTION:
Glaucoma can result in blindness if left untreated and as such it is extremely important to diagnose and treat the condition.

Usually doctors treat the first symptoms of glaucoma or ocular hypertension by prescribing eye drops. Unfortunately, there can be side effects associated with the use of these eye drops and there are reports of non-compliance due to difficulties in inserting these drops, all of which can impact on how effective this treatment regimen is.

The purpose of this study is to assess how well the new automated DSLT device for laser treatment of glaucoma or ocular hypertension works in comparison with the standard SLT and determine that it is as effective in reducing intraocular pressure.

DSLT or SLT will be performed in the study eye according to the randomization assignment. Eligible patients who sign the informed consent will be enrolled at each of the study sites, and undergo a washout (in the case of being medicated). After washout there will be a baseline visit, where continued eligibility is confirmed. Following confirmation of continued eligibility, 50% of patients being randomized to each treatment group. Randomization will be to a pre-determined randomization list.

The un-masked investigator(s) will open the envelope corresponding to the subject ID and administer the treatment as indicated by the randomization envelope. The masked ophthalmologist(s), who will perform the follow up, will be masked as to the nature of the treatment the patient underwent.

Only one eye per participant will be included in the study and they will be treated using either DSLT or SLT as per the randomized treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 years or older, with visual acuity > 6/60 in both eyes
2. Open angle glaucoma including exfoliative or pigmentary glaucoma or ocular hypertension
3. IOP ≥ 22mmHg to ≤35mmHg (after washout of any IOP-lowering medications)
4. Gonioscopically visible scleral spur for 360 degrees without indentation
5. Ability to visualize the peri-limbal sclera for 360 degrees (using a lid speculum)
6. Willing and able to participate in the 12-month study, to comply with the study procedures and to adhere to the follow-up schedule
7. Participant capable of giving informed consent

Exclusion Criteria:

1. Contraindications to conventional laser trabeculoplasty (e.g. corneal abnormalities, etc.)
2. Angle Closure Glaucoma
3. Congenital or developmental glaucoma
4. Secondary glaucoma except exfoliative or pigmentary glaucoma
5. Presence of any Peripheral Anterior Synechiae (PAS) in the study eye
6. Inability to conduct a reliable visual field (defined as fixation losses, false positives or false negatives greater than 33%)
7. Any of the following visual field findings using the Humphrey visual field analyzer the SITA-standard 24-2 program:

   1. A visual field MD of worse than -12dB
   2. Greater than or equal to 75% of points depressed below the 5% level and greater than or equal to 50% of points depressed below the 1% level on the PD plot
   3. At least 50% of points (i.e 2 or more) within the central 5 degrees with a sensitivity ≤0dB on the decibel plot
   4. Points within the central 5 degrees of fixation with a sensitivity <15 dB in both hemifields on the decibel plot
8. A visual field MD of worse than -12dB in the fellow eye
9. Cup:Disc Ratio of more than 0.8
10. More than three hypotensive mediations required
11. Prior incisional or laser glaucoma surgery (including previous SLT) in the study eye
12. Prior corneal refractive surgery
13. Complicated cataract surgery ≤ 6 months prior to enrollment
14. Presence of visually significant cataract in the opinion of the investigator
15. Clinically significant disease in either eye as determined by the Investigator
16. Clinically significant amblyopia in either eye
17. Dense pigmentation or haemorrhage in the peri-limbal conjunctiva or anterior sclera
18. Women who are pregnant or may become pregnant during the study
19. In the opinion of the investigator the participant might require other ocular surgery within the 12-month follow-up period, unless for further reduction of their IOP
20. Concurrent treatment with topical, nasal, inhaled or systemic steroids
21. Uncontrolled systemic disease that could impact the ability of the participant to attend follow up visits as per the discretion of the investigator
22. Participation in another clinical study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-22 (Actual)

PRIMARY OUTCOMES:
The difference between the two treatment groups between the mean baseline IOP and the mean IOP after the treatment | 6 months
  The mean baseline IOP (washed out for medicated patients) will be compared to the mean (washed out for medicated patients) IOP after the treatment

SECONDARY OUTCOMES:
Number of medications as compare to screening visit | 6 months
  Number of medications at 6 months as compared to screening/Visit 1 (before treatment) and compared between groups.
Proportion of subjects with at least 20% reduction in IOP from baseline | 6 months
  Proportion of subjects with at least 20% reduction in IOP at 6 months compared to baseline without surgical intervention

OTHER OUTCOMES:
Incidence of adverse events | 12 months
  Rates of Ocular Adverse events (AEs) in each treatment group at or prior to the 12 months visit

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Congdon, MD, MPH, Principal Investigator — Queens University Belfast
Locations (8):
- Israel (5):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
- Universita degli Studi di Genova, Genova, Italy
- United Kingdom (2):
  - Queens University Belfast, Belfast
  - Moorfields Eye Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gazzard G, Congdon N, Azuara-Blanco A, Blumenthal EZ, Gomelauri K, Zaliniyan M, Traverso CE, Bracha Z, Dvalishvili A, Solberg Y, Belkin M, Samuelson TW; GLAUrious Study Group. Randomized Noninferiority Trial of Direct Selective Laser Trabeculoplasty in Open-Angle Glaucoma and Ocular Hypertension: GLAUrious Study. Ophthalmology. 2025 Oct;132(10):1091-1104. doi: 10.1016/j.ophtha.2025.05.004. Epub 2025 May 9. PMID 40350086
- [Derived] Congdon N, Azuara-Blanco A, Solberg Y, Traverso CE, Iester M, Cutolo CA, Bagnis A, Aung T, Fudemberg SJ, Lindstrom R, Samuelson T, Singh K, Blumenthal EZ, Gazzard G; GLAUrious study group. Direct selective laser trabeculoplasty in open angle glaucoma study design: a multicentre, randomised, controlled, investigator-masked trial (GLAUrious). Br J Ophthalmol. 2023 Jan;107(1):62-65. doi: 10.1136/bjophthalmol-2021-319379. Epub 2021 Aug 25. PMID 34433548
- See also: Link to the manuscript in Ophthalmology — https://doi.org/10.1016/j.ophtha.2025.05.004